CLINICAL TRIAL: NCT03772080
Title: Early Education of Prematurity in High Risk Pregnancies-A Pilot Study
Brief Title: Prematurity Education in High Risk Pregnancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Rainbow Babies and Children's Hospital (Other)
Responsible Party: Principal Investigator, Rebecca Fish, Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20180789
Record Dates: First submitted 2018-11-01; First posted 2018-12-11 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Prematurity; High Risk Pregnancy
Keywords: Antenatal Counseling; Education
MeSH Terms: conditions — Premature Birth | interventions — Pregnancy, High-Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early counseling of prematurity in high-risk pregnancies (Experimental)
  Interventions: Other: Early counseling of prematurity in high-risk pregnancies.
- Standard counseling of prematurity in high-risk pregnancies (No Intervention)

INTERVENTIONS:
Other: Early counseling of prematurity in high-risk pregnancies. — Standardized information regarding prematurity, including associated complications and ways to decrease chances of preterm birth using web-based educational platform.
  Arms: Early counseling of prematurity in high-risk pregnancies

SUMMARY:
Prematurity is associated with significant morbidity and mortality. Given the high risk of death and disability, it is important for parents to understand the complications of prematurity so they can make decisions for their child. Unfortunately, these discussions often occur in the acute setting of threatened preterm labor when stress and anxiety make comprehension difficult. This study aims to improve parental understanding by providing early education of prematurity in the clinic setting for patients at high risk of preterm delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women between 22 0/7 and 34 6/7 weeks gestational age at high risk for premature delivery.

   1. Premature delivery defined as <37 0/7 weeks gestation.
   2. Any pregnant woman seen in the Maternal-Fetal Medicine Clinic deemed to be at high risk for premature delivery.
2. Pregnant women 16 years and older.
3. Pregnancy with singleton or twin gestation.
4. No major congenital malformation.
5. Women who are English speaking.

Exclusion Criteria:

1. Pregnant women <22 0/7 or >35 0/7 weeks gestational age.
2. Pregnant women less than 16 years old.
3. Multiple gestation greater than twins (triplets, quadruplets, etc).
4. Known major congenital malformation.
5. Women who are non-English speaking.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Parental knowledge of prematurity. | Outcome will be assessed on day 1 of the study. Data will be analyzed and reported at the completion of the study.
  Questionnaire to assess parental knowledge regarding basic concepts of prematurity, associated complications and factors that improve survival.
Parental satisfaction with prematurity education. | Outcome will be assessed on day 1 of the study. Data will be analyzed and reported at the completion of the study.
  Survey to assess usefulness of web-based educational tool and satisfaction with early education of prematurity.
Parental anxiety. | Outcome will be assessed on day 1 of the study. Data will be analyzed and reported at the completion of the study.
  Evaluation of parental anxiety associated with prematurity using validated six-item short-form of the Spielberger State-Trait Anxiety Inventory (STAI). The State-Trait Anxiety Inventory (STAI) measures presence and severity of anxiety. The inventory consists of two self-reporting subscales that evaluate the current state of anxiety (state anxiety subscale), as well as the propensity towards being anxious (trait anxiety subscale). The range for total score is 20-80, with a higher score indicating greater anxiety. The six-item version of the Spielberger State-Trait Anxiety Inventory (STAI: Y-6 item) is composed of three-questions from the original state anxiety subscale and three-questions from the original trait anxiety subscale. This shortened six-item inventory is a reliable and valid instrument when compared to the full forty-question inventory.

SECONDARY OUTCOMES:
Maternal compliance with maternal-fetal medicine provider follow up. | Outcome will be assessed up to 9 months following completion of the counseling intervention. Data will be analyzed and reported at the completion of the study.
  Frequency of no show and cancelled appointments during remainder of pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Fish, MD, Principal Investigator — UH, Cleveland Medical Center
Locations (1):
- UH Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No